CLINICAL TRIAL: NCT06343532
Title: Phase 1, Double-Blind, Placebo-Controlled, Parallel Group Study to Assess Potential Interactions Between Intravenous Cocaine and Oral SXC-2023
Brief Title: SXC-2023 Cocaine Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Promentis Pharmaceuticals, Inc. (Industry); Altasciences Company Inc. (Industry); Technical Resources International, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-SXC-Ph1b-001
Record Dates: First submitted 2024-03-13; First posted 2024-04-02 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Cocaine Use Disorder
Keywords: Cocaine; Benzoylecgonine; Glutamate; Cysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SXC-2023 (Experimental): SXC-2023: 800mg once a day for 7 days
  Interventions: Drug: SXC-2023
- SXC-2023 Placebo (Placebo Comparator): Placebo: 800mg once a day for 7 days
  Interventions: Drug: SXC-2023 Placebo

INTERVENTIONS:
Drug: SXC-2023 — 200 mg capsules
  Arms: SXC-2023
Drug: SXC-2023 Placebo — 200 mg capsules
  Arms: SXC-2023 Placebo

SUMMARY:
The goal of this clinical trial is to determine whether there are any interactions between the study drug and cocaine. Researchers will compare a treatment group and a placebo group to see if they experience any effects when administered cocaine after taking the treatment/placebo.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, parallel group study to compare the effects of SXC-2023 versus placebo control on intravenous cocaine's physiological and subjective effects in non-treatment seeking cocaine-experienced volunteers. Participants will be 18 to 59 years of age who have used cocaine by the smoked or intravenous route at least 6 times in the past 12 months prior to clinic intake, with at least one use within the past 3 months. Approximately twenty participants will be randomized to 2 groups, receiving either SXC-2023 or placebo treatment for 7 days. Adverse events and cardiovascular responses will be measured.

ELIGIBILITY:
Inclusion Criteria: In order to participate in the study, participants must:

1. Be participants who are cocaine-experienced and not seeking treatment for cocaine use disorder.
2. Males and females between 18 and 59 years of age, inclusive.

   • The masculine / feminine gender is used without any discrimination and with the aim to lighten the text.
3. Have a body mass index (BMI) within a range of 17.0 to 36.0 kg/m2 and a minimum weight of at least 50.0 kg at screening.
4. Have experience using cocaine by the smoked or i.v. route at least 6 times over the participant's lifetime prior to clinic intake (Day -3) and at least one use within the past 3 months.
5. Provide a urine sample positive for cocaine at least once during screening (Days -28 to -4) and a urine test negative for cocaine at clinic intake.
6. Be able to verbalize understanding of consent form, able to provide written informed consent, and verbalize willingness to complete study procedures.
7. A female study participant must meet one of the following criteria:

   * If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 30 days prior to the first administration of the study medication, during the study, and for at least 30 days after the last dose of the study medication. An acceptable method of contraception includes one of the following:

     i. Abstinence from heterosexual intercourse ii. Hormonal contraceptives (oral/injectable/implant/insertable hormonal birth control products, transdermal patch) iii. Intrauterine device (with or without hormones) OR agrees to use a double barrier method (e.g., condom and spermicide) during the study and for at least 30 days after the last dose of the study medication.
   * If a female of non-childbearing potential - should be surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion) or in a menopausal state (at least 1 year without menses), as confirmed by FSH levels (≥ 40 mIU/mL).

   A male study participant that engages in sexual activity that has the risk of pregnancy must agree to use a double barrier method (e.g., condom and spermicide) and agree to not donate sperm during the study and for at least 90 days after the last dose of the study medication.
8. Be able to comply with protocol requirements, rules and regulations of the study site, and be likely to complete all the study treatments.

Exclusion Criteria: In order to participate in the study, participants must not:

1. Have a current or past history of seizure disorder, including alcohol- or stimulant-related seizure, febrile seizure, or significant family history of idiopathic seizure disorder.
2. Have any previous medically adverse reaction to cocaine, including loss of consciousness, chest pain, paranoid reaction or seizure.
3. Have clinically significant findings in the opinion of an investigator based on the MINI (version 7.0) neuropsychiatric interview.
4. Be pregnant or lactating.
5. Have a sitting systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg and heart rate > 100 beats per minute at screening and clinic intake.
6. Have a history of liver disease or current elevation of aspartate aminotransferase (AST), alanine aminotransferase (ALT), 2 × the upper limit of normal.
7. Blood donation (excluding plasma donation) of approximately 500 mL within 56 days prior to screening.
8. Plasma donation within 7 days prior to screening.
9. Treatment with an investigational drug within 30 days or 5 times the half-life (whichever is longer) prior to screening.
10. Have any clinically significant finding on medical history, physical examination, clinical laboratory test, vital signs or ECGs that contraindicate participation in the study.
11. Have a history of suicide attempts or current or recent evidence of suicidal ideation in the past 12 months based on the Columbia-Suicide Severity Rating Scale (C-SSRS).
12. Have a positive urine drug screen upon clinic intake (Day -3) for any of the following drugs: alcohol, amphetamine/methamphetamine, barbiturates, benzodiazepines, buprenorphine, cocaine, fentanyl, 3,4-methylenedioxymethamphetamine (MDMA), methadone, phencyclidine/phenylcyclohexyl piperidine (PCP), propoxyphene, and opioids (e.g., codeine, heroin, morphine, oxycodone, etc.). If a participant presents with a positive urine drug screen for cocaine or alcohol at clinic intake (Day -3), the participant may be rescheduled one time at the discretion of an investigator or designee as long as clinic intake is within the total screening window.
13. Have used any prescription drugs within 14 days of clinic intake or non-prescription drugs or herbal remedies within 7 days of clinic intake.
14. Be unable to distinguish between a 20 mg and 40 mg dose of cocaine i.v. based on the high effects VAS at either the 5 or 10 minute time point during the screening infusion.
15. Have a positive serology for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCVab), or human immunodeficiency virus (HIV).
16. Have positive results for a coronavirus disease 2019 (COVID-19) test performed after screening is complete and participant is confirmed, but prior to admission.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) of Oral SXC-2023 Co-administered with Intravenous Cocaine | Study Days -2,1,2,8,9,11
  Determine if there are significant interactions between oral SXC-2023 treatment concurrent with 20 and 40 mg intravenous cocaine infusions by measuring incidence of treatment emergent adverse events using the most recent version of the Medical Dictionary of Regulatory Activities (MedDRA) preferred terms, relationship to the treatment, and maximum severity, either reported by the subject or by clinically significant abnormal findings on:
  i. Physical examination ii. Rate of change in vital signs assessments of heart rate, blood pressure, respiration rate, and temperature iii. Rate of change in ECG assessment iv. Rate of clinical laboratory changes

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Principal Investigator — Altasciences Clinical Kansas, Inc.
Locations (1):
- Altasciences Clinical Kansas, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided